CLINICAL TRIAL: NCT05170178
Title: Cracking the Code of Crying Babies: How Familiarity Changes the Interpretation of Cries
Acronym: BEBEDOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21CH161; ANSM (Other: 2021-A02270-41)
Record Dates: First submitted 2021-12-22; First posted 2021-12-27 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-06

CONDITIONS: Magnetic Resonance Imaging; Neuronal Activity
Keywords: baby cries; pain; brain responses; fmRI; familiarity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Group with parental experience caring for infants (20 men and 20 women) Group with professional experience in caring for infants (20 women)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Women with parental experience caring for infants (Experimental): Women parent of a child under 2 years old
  Interventions: Behavioral: inclusion and familiarization; Behavioral: fMRI acquisition and closure
- Men with parental experience caring for infants (Experimental): Men parent of a child under 2 years old
  Interventions: Behavioral: inclusion and familiarization; Behavioral: fMRI acquisition and closure
- Women with professional experience in caring for infants (Experimental): Women in daily contact with infants in professional circle (e.g., nannies, pediatricians, midwives, maternity nurses) without dependent children under 2 years old
  Interventions: Behavioral: inclusion and familiarization; Behavioral: fMRI acquisition and closure

INTERVENTIONS:
Behavioral: inclusion and familiarization — * presentation of the study purpose and the protocol to the volunteer
  * clinical examination to check inclusion and exclusion criteria
  * Familiarization with the crying of one assigned baby, by listening to several bath cries from this baby
Behavioral: fMRI acquisition and closure — * Second phase of familiarization, listening again to bath cries of "their" assigned baby. These cries will be different from those listened during the first familiarization phase.
  * MRI acquisition: after acquisition of the anatomical images (5 min), the subjects will listen to 64 cries divided into 4 functional MRI sessions of 10 minutes each. The cries will be those of "their" baby or of unknown babies, evoked in a painful (vaccination) or a non-painful (bath) situation, presented in a pseudo-random order. Participants will be asked to assess whether they recognize "their" baby (yes/no) and whether they recognize a pain cry (yes/no).
  * debriefing
  * Protocol ending

SUMMARY:
Understanding babies' signals is essential to meet their needs. Recent works suggest that crying provides useful information, not only allowing parents to recognize their baby among others (static information), but also to distinguish between mild discomfort and pain cries (dynamic information). The perception of this information by adults involves a "parental" brain network including brain areas involved in empathy, attention, emotional regulation, motor as well as regions of the limbic system or associated with the reward network.

DETAILED DESCRIPTION:
This network is involved when listening to cries of familiar babies, or pain cries. How do we become specialist of a baby's cries? To date, no functional imaging study has examined the specific brain activations when listening to the cries of a familiar baby in different situations, particularly painful ones.

ELIGIBILITY:
Inclusion Criteria

For all volunteers:

* Affiliated or entitled to a social security plan
* Right-handed by the Edinburgh laterality test
* Having given free, informed and written consent to participate in the study
* Having given their consent for the communication of the MRI results to their attending physician

Group with parental experience caring for infants :

* Men or women between 18 and 50 years old
* Parent of a child under 2 years old

Group with professional experience in caring for infants

* Women between 18 and 50 years old
* Without dependent children under 2 years of age
* People in daily contact with infants in the professional circle (e.g. nurses, pediatricians, midwives, maternity nurses, etc)

Exclusion Criteria

* Pregnant women, parturient, nursing mothers or parents
* Persons deprived of liberty, hospitalized without consent, hospitalized for purposes other than research
* Minors
* Adults under legal protection (guardianship) or unable to express their consent
* Subjects with contraindications to the MRI examination: use of a pacemaker or an insulin pump, wearing a metallic prothesis, an intracerebral clip or a piercing, claustrophobia,
* Taking medication for less than 12 hours,
* Neurological, psychiatric or auditory history or deficits.
* Anxiety and/or depressive disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
BOLD signal (blood oxygen level-dependent) | during the whole listening session
  Measurement of the BOLD signal by fMRI (functional magnetic resonance imaging) in adults during listening to natural cries of a familiar baby and unknown babies, in two painful (vaccination) or non-painful (bath) situations.

SECONDARY OUTCOMES:
participants'experience at caring for babies | At the inclusion visit
  Experience at caring for babies : Yes or No
participants' sex | At the inclusion visit
  Sex : Male or female

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (2):
- France (2):
  - HCL, Bron
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No